CLINICAL TRIAL: NCT04887597
Title: EBIO - Enthesitis Biopsy Study
Acronym: EBIO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EBIO
Record Dates: First submitted 2019-09-25; First posted 2021-05-14 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-05

CONDITIONS: Psoriatic Arthritis; Enthesitis; Biopsy
Keywords: Enthesitis; Imaging; Psoriatic Arthritis; Biopsy
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This is an open label interventional study in 10 patients with enthesitis in psoriasis arthritis (PsA). The study is composed of a single arm receiving secukinumab for the duration of 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Secukinumab Treatment (Experimental): all patients receive Secukinumab as well as a biopsy before and after treatment
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — The study is composed of a single arm receiving secukinumab for the duration of 6 months.

SUMMARY:
The purpose of this Phase IV study is to determine the effect of secukinumab on total immune cell numbers obtaines by entheseal biopsy in the inflamed human entheses in patients with Psoriatic Arthritis. This is a single arm, single centre, prospective, open label study with secukinumab.

DETAILED DESCRIPTION:
Psoriatic arthritis (PsA) is a heterogeneous inflammatory rheumatologic disorder characterized by inflammatory arthritis, enthesitis, dactylitis and spondylitis, affecting 6% to 39% of the patients suffering from psoriasis. The exact prevalence of PsA is unknown. Estimates of incidence vary from 0.3% to 1% of the population. Disease onset typically occurs between the ages of 30 and 55 years, and affects both genders equally. PsA is classified as a seronegative spondyloarthropathy (SpA) because it shares certain features with other conditions included in that group. Indeed, spinal involvement has been reported in approximately 50% of patients with PsA. In addition, PsA is associated with enthesitis and dactylitis, which are extra-articular features common to SpA. Finally, the majority of patients with PsA are negative for the rheumatoid factor. Recent studies have challenged the assertion that PsA is a more benign disease than rheumatoid arthritis. There is an increasing body of evidence that suggests that PsA patients experience progressive joint destruction over a relatively short period of time. The results from these studies indicate that PsA is erosive and deforming in nearly half of the patients, with joint damage appearing in the first years of disease onset. Other investigators later confirmed that 41% of the patients developed erosive disease within 2 years of onset of symptoms.

Diagnosis and treatment as early as possible has become the standard of care in rheumatoid arthritis in order to prevent disease progression, irreversible functional impairment and premature death. Since the 1970s, it has also been recognized that each inflammatory lesion (joint synovitis, tenosynovitis, dactylitis, enthesitis, sacroiliitis, and spondylitis) can develop without symptoms or signs that are recognizable by the patient and the physician. Such patients can be considered to have subclinical or "occult" PsA. Support for this notion comes from imaging studies providing evidence for the existence of subclinical inflammatory changes in patients with psoriatic skin disease using MRI or high-resolution ultrasound scans.

The investigators focused on the concept of "pre-clinical" changes in their own observational study. Patients suffering from psoriasis with no present or past signs of joint manifestations to stringently rule out clinical joint involvement, have been investigated. The investigators recently described that patients with psoriasis, but without PsA, exhibit entheseophytes as the result of pathological bone formation in the joints as a pathological hallmark of PsA. Recent work has identified enthesial pathology as a specific part of the PsA disease process. Entheses may represent the primary site of musculoskeletal changes in psoriasis patients developing PsA. In particular, the understanding of enthesial structures as an organ with a high degree of structural and functional organisation and the coining of the term 'synovio-entheseal complex' have extended the view on PsA. These concepts are of potential importance in searching for the discrete changes of the joints in patients with psoriatic skin disease. This finding reinforces the pathophysiological role of the entheses in patients with psoriatic disease. Apparently, enthesial changes can occur in the sole presence of skin disease and do not require the clinical arthritis corroborating the concept of an intrinsic clinical connection between the skin and the entheses, which has been previously suggested by molecular studies referring to the role of interleukin-23 as a linker between skin and enthesial pathology.

In the peripheral joints, entheses can be found at the attachment of the collateral ligaments and the circumferential insertion of the capsule itself, which are also known as 'synovio-entheseal complexes' and are highly prone to structural bone changes. Furthermore, functional entheses exist at the dorsal and palmar sites of the MCHs serving as pulleys for the extensor and flexor tendons, respectively. Importantly, these mechanically exposed locations were identical with the sites of new bone formation, suggesting a tight connection between mechanical factors and the bone response observed in psoriasis patients.

Findings provide new evidence for the existence of a Deep Koebner Phenomenon at the enthesial sites in psoriasis patients. In its original description, this phenomenon corresponds to the trigger of inflammation and acro-osteolysis by a discrete traumatic injury. New findings extend the concept of the Deep Koebner Phenomenon suggesting a pathological tissue response to mechanical stress in psoriasis patients. This response affects the mechanically exposed sites of the body, which are the skin and the entheses. The specific importance of entheseophyte formation in psoriasis patients is also supported by the observation that the burden of bone erosions was not significantly enhanced in psoriasis patients compared with healthy controls.

Moreover enthesitis is a frequent manifestation in PsA and SpA. Dependent on studies between 23% and 70% of patients with PsA/SpA show enthesitis. Enthesitis is characterized by inflammation at specific anatomical sites, where ligaments, tendons and joint capsules attach to bone. The main clinical manifestations of enthesitis is pain while swelling is infrequent. Pain can be severe, persistent and resistent to treatment.

Up-to-date no synovial or enthesial tissue biomarkers are available to stratify treatment strategies in regard to an anti-inflammatory response to bDMARD therapies in active psoriatic arthritis with enthesitis. Looking at other medical disciplines such as the oncology field, where detailed histological, immunohistochemical and even genetic analysis of tumor tissue for a personalized diagnostic, therapeutic and prognostic decision are performed, in rheumatology (inflammatory discipline) we are still far from a personalized diagnostic, therapeutic and prognostic approach based on tissue biomarker to better help and advice patients. Fortunately, a growing variety of medications such as bDMARDs are available, however investigators are still in a "try and error" situation.

Obtaining and analyzing enthesial tissue biopsies prior and after treatment with an anti-IL17 monoclonal antibody (secukinumab) might allow the investigators to identify biomarkers for treatment responses, using histological, immunohistochemical, molecular and flow cytometry techniques to further add information to the understanding of inflammation and entheses repair processes.

Virtually all information on enthesitis to date is based on either preclinical models or the clinical assessment of tender points in humans creating a huge unmet need for a better understanding of human enthesitis. To date only one single biopsy study of enthesitis has been carried out, which assessed acute enthesiopathy in peripheral SpA patients. In light of the availability of drugs with high clinical efficacy on enthesitis, such as IL-17 blockers, and the preclinical evidence for a role of the IL-23/IL-17 pathway in enthesitis, human studies are needed to assess how and to what extent IL-17 inhibition ameliorates enthesitis. Serum studies can hardly replace biopsy studies in this respect, since many of the processes in enthesitis are local.

Based on this situation the investigators propose a combined biopsy-imaging study in patients with PsA with active clinical enthesitis of the lateral epicondyle of the humerus or achilles tendon. Patients will receive a 6-month treatment with secukinumab and the effect on enthesial inflammation will be assessed by histology and mRNA assessment as well as combined imaging.

ELIGIBILITY:
The trial population consists of patients of both sexes, aged ≥ 18 years, with active psoriatic arthritis and an indication for systemic treatment.

Patient eligible for study participation will have to fulfil the following requirements:

* Must be male or female and aged > 18 years at time of consent
* Clinical signs of enthesitis for at least 6 weeks prior to enrolment
* Indication for systemic treatment for PsA according to guidelines
* Patients who failed to respond to or who have a contraindication to, or are intolerant to other systemic therapy including cyclosporine or methotrexate
* bDMARD and tsDMARD naive
* Must understand and voluntarily sign an informed consent form including written consent for data protection
* Must be able to adhere to the study visit schedule and other protocol requirements
* Male subjects (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with Females of Childbearing Potential (FCBP) while on study medication and for at least 28 days after taking the last dose of study medication.
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening and must be willing to use one effective form of birth control when engaging in reproductive sexual activity while on study medication and for at least 28 days after taking the last dose of study medication.

Effective contraception methods include:

1. Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception;
2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy);
3. total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment;
4. Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner of that Patient;
5. Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical/vault caps)
6. Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1 percent), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS); In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking investigational drug; In case local regulations deviate from the methods listed, local regulations apply and will be described in the ICF; Women are considered post-menopausal and not of child bearing potential if they have had at least 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago.

Additional eligibility criterium prior to enthesial biopsy:

- Presence of inflammation (enthesitis, synovitis, tendinitis, osteitis or tenosynovitis) in MRI or ultrasound examination of the elbow/ankle must be detectable

Exclusion criteria:

* Any contraindications for the treatment with secukinumab
* Subjects requiring systemic anticoagulation therapy or suffering from coagulation disorders or any other condition which might interfere with enthesitis tissue sampling
* IBD (e.g. Crohn´s disease, ulcerative colitis)
* Investigational study drug within 4 weeks (or 5 half-lives, whichever is longer) prior to enrolment
* Patients taking high-potency opioid analgesics, including but not limited to, methadone, hydromorphone, and morphine
* Any contraindication or unwillingness to perform MRI
* Rheumatologic, inflammatory diseases, including but not limited to: AS, RA
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception
* Any underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, psychiatric, endocrine, cardiac, infectious or gastrointestinal conditions which in the opinion of the investigator immune-compromises the patient and/or places the patient at unacceptable risk for participation in a secukinumab therapy
* Active systemic infections during the last two weeks (exception: common cold) prior to enrolment.
* Evidence of tuberculosis infection as defined by either a positive purified protein derivative (PPD) skin test (the size of induration will be measured after 48-72 hours, and a positive result is defined as an induration of ≥ 5mm or according to local practice/guidelines), or a positive Quantiferon test. Patients with a positive test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the patient has no evidence of active tuberculosis. If presence of latent tuberculosis is established then treatment according to local country guidelines must have been initiated prior to enrolment.
* Infection with human immunodeficiency virus (HIV) Hepatitis B (HBV) or Hepatitis C (HCV)
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system (except for basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed), treated or untreated within the past 5 years prior to enrolment.
* History or evidence of ongoing alcohol or drug abuse, within the last six months prior to enrolment.
* Planned administration of live vaccines during the study period or within 6 weeks prior to enrolment.
* Patients who possibly are dependent on the Sponsor, the Principal Investigator or Investigator (e.g. family members).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Percent of patients with reduction of total immune cell (PMN, M, T cells, B cells, ILC3, Mast cells) numbers by at least 50 percent in the enthesial tissue after 24 weeks of treatment with secukinumab | baseline and 6 months
  To define the effect of IL-17A inhibition on total immune cell numbers (PMN, M, T cells, B cells, ILC3, Mast cells) in the inflamed human entheses.

SECONDARY OUTCOMES:
Change in numbers of MPO+ neutrophils and CD11b+ positive macrophages in enthesial biopsies | baseline and 6 months
  To define the effect of IL-17A inhibition on the numbers of IL-17 expressing cells in the inflamed human entheses and the expression of IL-17 pathway and bone formation genes in the inflamed human entheses
Enthesitis and osteitis in MRI (elbow/ankle) (yes/no) | baseline and 6 months
  To define the effect of IL-17A inhibition onthe expression of IL-17 pathway and bone formation genes in the inflamed human entheses
Enthesitis in ultrasound examination (elbow/ankle) (yes/no) greyscale and doppler | baseline and 6 months
  To define the effect of IL-17A inhibition onthe expression of IL-17 pathway and bone formation genes in the inflamed human entheses
Change in clinical enthesitis (SPARCC,LEI,MASES) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Change in clinical arthritis (SJC;TJC; DAPSA) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Change in clinical skin disease (PASI) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Number of subjects with minimal disease activity (MDA) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Change in Pain (VAS) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Change in Physical function (HAQ-DI) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality
Change in Impact of disease (PSAID) | baseline and 6 months
  To define the effect of IL-17A inhibition on clinical signs of enthesitis, arthritis, skin disease, physical function and life quality

CONTACTS AND LOCATIONS:
Overall Officials: Markus Neurath, Prof, Study Chair — Dean University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Department of Internal Medicine 3, Rheumatology and Immunology, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No